CLINICAL TRIAL: NCT01287975
Title: ARTS-BCI: Advanced Brain Computer Interface (BCI) Technology for Wrist and Hand Rehabilitation After Stroke
Brief Title: Brain Computer Interface (BCI) Technology for Stroke Hand Rehabilitation
Acronym: ARTS-BCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Institute for Infocomm Research (Other)
Responsible Party: Principal Investigator, Chua Sui Geok, Karen, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SERC Grant No: 092 148 0066
Record Dates: First submitted 2011-01-26; First posted 2011-02-02 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Brain Computer Interface; Upper Limb Rehabilitation; EEG-based Motor Imagery; Robotic Rehabilitation; Haptic Knob
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Occupational Therapy (Active Comparator): Standard Occupational Therapy for Wrist and Hand Training
  Interventions: Other: Occupational Therapy
- BCI Haptic Knob (Experimental): BCI controlled robotic-assisted training for wrist and hand
  Interventions: Device: BCI Haptic Knob
- Haptic Knob (Experimental): Robotic-assisted training for wrist and hand
  Interventions: Device: Haptic Knob

INTERVENTIONS:
Other: Occupational Therapy — Use of conventional manual facilitation and function-based training used in conventional occupational therapy training for post-stroke upper limb weakness.
  Training is modelled along the neurodevelopmental techniques and will include stretching, tone management, weight bearing exercises, movement facilitation, selfcare training, arm ergometry by arm bicycles and grip strength training.
  Training intensity is 1.5 hours for 3 times a week for 6 weeks consecutively.
  Arms: Standard Occupational Therapy
Device: BCI Haptic Knob — BCI based robotic rehabilitation works by detecting the motor intent of the user from electroencephalogram signals to drive the robotic rehabilitation via Haptic Knob. Training intensity is 1.5 hours for 3 times a week for 6 weeks consecutively.
  Arms: BCI Haptic Knob
Device: Haptic Knob — Haptic Knob is an upper limb robot designed for use in robotic-assisted rehabilitation of the stroke wrist and hand. Training intensity is 1.5 hours for 3 times a week for 6 weeks consecutively.
  Arms: Haptic Knob

SUMMARY:
This study is carried out to find out if Brain Computer Interface (BCI) technology or BCI technology coupled with robotic technology using a Haptic Knob will benefit patients with arm paralysis after stroke. BCI uses EEG-based motor imagery to detect user's thinking abilities which control motor movement. Haptic Knob is a novel robotic device, which specifically trains the wrist and hand with intensive repetitions in a supported environment.

DETAILED DESCRIPTION:
Physical therapy approaches are the de facto rehabilitation for stroke, which involve human therapists to assist stroke patients in recovering their motor ability. Modern rehabilitation technologies include robotics, functional electrical stimulation, transcranial magnetic stimulation and virtual reality. Robotic rehabilitation alleviates the labor-intensive aspects of physical rehabilitation by human therapists and could potentially improve the productivity of stroke rehabilitation. However, it is fundamentally based on movement repetition with visual feedback that helps stroke patients improve motor ability in their weak stroke-affected arms and legs. However, the robot is still able to move the weak part of the patient even if the patient is not attentive towards the training and thus the robotic training becomes a passive activity. In contrast, BCI-based robotic training works by ensuring active engagement by the hemiparetic patients in making a volitional movement. In addition, hemiplegic or locked-in stroke patients who do not have any motor power on the affected limbs are then able to engage and perform a volitional movement on these affected limbs.

BCI-based robotic rehabilitation fills this gap by detecting the motor intent of hemiplegic patients from the Electroencephalogram (EEG) signals to drive the robotic rehabilitation. This BCI-based robotic rehabilitation for stroke research project was jointly conducted by Tan Tock Seng Hospital (TTSH), National Neuroscience Institute (NNI) and Institute for Infocomm Research (I2R). Preliminary clinical trials performed at TTSH have shown that stroke patients can operate the BCI as effective as healthy subjects.

Specifically, this research project will address the following gaps in the area of rehabilitation for stroke:

1. Single-modal BCI - The current system employs a single modal non-invasive EEG-based BCI that detects motor intent using at least 2.5 seconds of EEG data. Hence, the research of an advanced multi-modal BCI such as synergizing near-infrared spectroscopy with EEG to yield a more responsive and effective BCI-based robotic rehabilitation system is proposed.
2. Standard therapy - The current system employs a standard therapy for all the stroke patients. However, physiotherapists and occupational therapists usually adopt a more individualized therapy for each stroke patients. Hence, research on an individualized therapy for each stroke patient according to his or her learning rate and neurological insult is proposed.
3. Only physiological rehabilitation - The current system only performs physiological rehabilitation of motor functions of stroke patients. Currently some validated scales for post-stroke depression such as Beck depression inventory, CES-D, Zung scale, State trait, HADS etc are difficult to administer in stroke patients who cannot participate with assessment due to impaired language or cognitive abilities. Hence an advanced BCI-based rehabilitation system that also detects the mental state of the stroke patient is proposed to cover both physiological and psychological rehabilitation.
4. Upper Limb rehabilitation - The current system which uses the clinically-proven MIT Manus robotic rehabilitation system, only performs upper limb rehabilitation for stroke patients in gross reach patterns. Human hand skills, in contrast, consist of more complex manipulation movement patterns which can be intervened by BCI-based robotic rehabilitation. Hence, an advanced BCI-based rehabilitation system that covers the hand function is proposed to cover the rehabilitation of the entire upper extremity.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21-80 years with first-ever clinical stroke, within 1-24 months onset.
2. Stroke type: ischemic or haemorhagic.
3. Fugl-Meyer motor score of the upper limb range from 10-50 or
4. Motor power MRC grade 3-5 in shoulder abductors and elbow flexors, and 0-3 in wrist dorsiflexors and finger flexors
5. Ability to pay attention and maintain supported sitting for 1 hour continuously.
6. Able to give own consent and understand simple instructions
7. Fulfills BCI and Haptic knob physical screening trial.

Exclusion Criteria:

1. Functional status: severe aphasia or inattention, unstable medical conditions which may affect participation (e.g. unresolved sepsis, postural hypotension, end stage renal failure) or anticipated life expectancy of <1 year due to malignancy or neurodegenerative disorder)
2. Hemispatial neglect (visual or sensory) or severe visual impairment despite visual aids.
3. Epilepsy, severe depression or psychiatric disorder.
4. Recurrent stroke
5. Skull defect as this would affect physical fit of EEG cap interface.
6. Local arm factors: Severe spasticity Modified Ashworth scale >2 in any region, visual analogue scale (VAS score) >4/10, fixed joint contracture , patients with poor skin conditions, infections or eczema which may potentially be worsened by robotic shell contact.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Measures the change of upper limb motor function post-stroke
Fugl Myer Upper Limb Motor Assessment | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Measures changes in post-stroke upper limb movement

SECONDARY OUTCOMES:
Frenchay Arm Test | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  To measure performance in functional hand use post stroke
Grip Strength | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Use of grip dynamometer to measure changes in grip strength
Modified Ashworth Scale | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Measure changes in spasticity of the affected limb
Functional Independence Measure (Motor) | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Measures participation in activities of daily living.
Pain Score | Measurements at 2 weeks prior to intervention, just before start of intervention, at midpoint of intervention, at completion of intervention, at 3 months post intervention and at 6 months post-intervetion
  Use of visual analogue scale of 0-10 for pain measurement

CONTACTS AND LOCATIONS:
Overall Officials: Karen SG Chua, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

REFERENCES:
- [Background] Ang KK, Guan C, Chua KS, Ang BT, Kuah C, Wang C, Phua KS, Chin ZY, Zhang H. Clinical study of neurorehabilitation in stroke using EEG-based motor imagery brain-computer interface with robotic feedback. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:5549-52. doi: 10.1109/IEMBS.2010.5626782. PMID 21096475
- [Background] Arvaneh M, Guan C, Ang KK, Ward TE, Chua KSG, Kuah CWK, Ephraim Joseph GJ, Phua KS, Wang C. Facilitating motor imagery-based brain-computer interface for stroke patients using passive movement. Neural Comput Appl. 2017;28(11):3259-3272. doi: 10.1007/s00521-016-2234-7. Epub 2016 Mar 4. PMID 29051688
- [Background] Ang KK, Guan C, Phua KS, Wang C, Zhou L, Tang KY, Ephraim Joseph GJ, Kuah CW, Chua KS. Brain-computer interface-based robotic end effector system for wrist and hand rehabilitation: results of a three-armed randomized controlled trial for chronic stroke. Front Neuroeng. 2014 Jul 29;7:30. doi: 10.3389/fneng.2014.00030. eCollection 2014. PMID 25120465
- [Background] Ang KK, Guan C, Chua KS, Phua KS, Wang C, Chin ZY, Zhou L, Tang KY, Joseph GJ, Kuah C. A clinical study of motor imagery BCI performance in stroke by including calibration data from passive movement. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6603-6. doi: 10.1109/EMBC.2013.6611069. PMID 24111256